CLINICAL TRIAL: NCT01456026
Title: Acute Effects of Food Advanced Glycation Endproducts on Macrovascular Function in Subjects With Type 2 Diabetes Mellitus
Brief Title: Effects of Food Advanced Glycation Endproducts on Vascular Function in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: Heart and Diabetes Center North-Rhine Westfalia (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Exogene-AGE
Record Dates: First submitted 2011-10-14; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Advanced glycation endproducts; Endothelium
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glycated beta-lactoglobulins (Experimental): In this randomized, double blind,cross-over study, half of the subjects will receive on one day a beverage with a high AGE content and will be switched after a wash-out of min. 7 days to receive a low-AGE beverage (comparator). The other half will receive the beverages in inverse sequence.
  Interventions: Dietary Supplement: Glycated beta-lactoglobulins.
- Non-glycated beta-lactoglobulins (Active Comparator): In this randomized, double blind,cross-over study, half of the subjects will receive on one day a beverage with a high AGE content and will be switched after a wash-out of min. 7 days to receive a low-AGE beverage (comparator). The other half will receive the beverages in inverse sequence.
  Interventions: Dietary Supplement: Non-glycated beta-lactoglobulins

INTERVENTIONS:
Dietary Supplement: Glycated beta-lactoglobulins. — oral, 20 g, single administration
  Arms: Glycated beta-lactoglobulins
Dietary Supplement: Non-glycated beta-lactoglobulins — 20 g, oral, single administration,
  Arms: Non-glycated beta-lactoglobulins

SUMMARY:
Recent evidence supports detrimental effects of advanced glycation endproducts (AGE) on vascular function (VF). Though, the effect of AGE-modified proteins alone on vascular function remained unknown. Therefore, the aim of our study is to investigate the effects of heat-treated, glycated beta-lactoglobulins (BLG) on vascular function in subjects with type 2 diabetes mellitus (T2DM) and to compare it to non-glycated, heat-treated BLG.

DETAILED DESCRIPTION:
In a double-blind, controlled, randomized, cross-over manner, 19 subjects with T2DM will receive on 2 different days beverages containing either glycated, heat-treated BLG or non-glycated, heat-treated BLG.

Macrovascular (brachial ultrasound of flow mediated dilatation -FMD) and microvascular function (laser-doppler measurements of reactive hyperemia at the hand) at baseline (T0), as well as 90 (T90) and 180 (T180) minutes after each beverage will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus

Exclusion Criteria:

* Other types of diabetes
* Major cardiovascular complications within 6 months prior to screening
* Major diabetes complications
* Failure to give informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Postprandial Change from Baseline in Flow Mediated Dilatation | Baseline, 90 and 180 min after oral intake of food AGE
  Macrovascular (brachial ultrasound of flow mediated dilatation -FMD) will be measured at baseline (T0), as well as 90 (T90) and 180 (T180) minutes after each beverage. The hypothesis of our study is that an AGE-rich beverage acutely impairs FMD more than a beverage with a low AGE content.

SECONDARY OUTCOMES:
Postprandial Change from Baseline in Microcirculation (Laser-Doppler measurements of reactive hyperemia at the hand) | Baseline, 90 and 180 min. following food AGE intake.
  Microvascular function will be measured at baseline (T0), as well as 90 (T90) and 180 (T180) minutes after each beverage. The hypothesis of our study is that an AGE-rich beverage acutely impairs microvascular function more than a beverage with a low AGE content.

CONTACTS AND LOCATIONS:
Overall Officials: Alin O Stirban, M.D., Principal Investigator — Profil Institute for Metabolic Research GmbH
Locations (1):
- Heart and Diabetes Center North-Rhine Westfalia, Bad Oeynhausen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Stirban A, Kotsi P, Franke K, Strijowski U, Cai W, Gotting C, Tschoepe D. Acute macrovascular dysfunction in patients with type 2 diabetes induced by ingestion of advanced glycated beta-lactoglobulins. Diabetes Care. 2013 May;36(5):1278-82. doi: 10.2337/dc12-1489. Epub 2012 Dec 13. PMID 23238657